CLINICAL TRIAL: NCT06069479
Title: Comparing Effectiveness of a Conservative Policy to Craniofacial Surgery in Children With Trigonocephaly: an Observational Cohort Study on Clinical Outcomes, Psychosocial Wellbeing, and Costs
Brief Title: Comparing Conservative to Surgical Treatment of Trigonocephaly Craniofacial Surgery in Children With Trigonocephaly: an Observational Cohort Study on Clinical Outcomes, Psychosocial Wellbeing, and Costs
Acronym: Treat Trigono
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: LAPOSA (Unknown); IJsselland ziekenhuis (Unknown); Sint Franciscus Gasthuis (Other)
Responsible Party: Principal Investigator, Irene Mathijssen, prof.dr. MBA-H, Erasmus Medical Center
Other Study IDs: PaNaMaID 9517
Record Dates: First submitted 2023-10-02; First posted 2023-10-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-01

CONDITIONS: Metopic Synostosis
MeSH Terms: conditions — Craniosynostoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Conservative group: Children with trigonocephaly that are treated conservatively.
- Surgical group: Children with trigonocephaly that are treated surgically.
  Interventions: Procedure: craniofacial surgery

INTERVENTIONS:
Procedure: craniofacial surgery — Surgical treatment, either stripcraniectomy or fronto-orbital advancement
  Groups: Surgical group

SUMMARY:
RESEARCH QUESTION Is the effectiveness of conservative policy comparable to that of surgery in children with trigonocephaly, with regard to clinical outcomes and psychosocial functioning, stress for parents, and costs? DESIGN Observational cohort study in children, aged 0 to 8 years old, with trigonocephaly, excluding metopic ridging (physiologic early closure of metopic suture), treated conservatively or surgically.

OUTCOME MEASURES Primary: Head growth decline, indicating raised intracranial pressure Secondary: fundoscopy, cognition, behavior, refraction and vision, forehead shape, quality of life, posttraumatic stress, decisional conflict, costs.

DETAILED DESCRIPTION:
HYPOTHESIS Conservative treatment is non-inferior to surgery with regard to clinical outcomes, causes less burden of disease, and is cost-effective.

STUDY DESIGN Observational cohort study STUDY POPULATION Children, aged 0 to 8 years old, with trigonocephaly, excluding metopic ridging (physiologic early closure of metopic suture) INTERVENTION Conservative policy USUAL CARE/COMPARISON Craniofacial surgery OUTCOME MEASURES Primary: Head growth decline (head circumference in SD), indicating raised intracranial pressure Secondary: fundoscopy, cognition, behavior, refraction and vision, forehead shape, quality of life, posttraumatic stress, decisional conflict, costs. Repeated measures at 0, 2, 4, 6, 8 years of age SAMPLE SIZE/DATA ANALYSIS Eligible patients <= 3 years of age are included since Sept 2022 Sample size 440 patients <1 year of age: 195 surgery and 245 conservative

Non-inferiority with regard to head growth from 0-4 years (annual measurement) is determined using a linear mixed model adjusted for confounders:

severity of phenotype, sex, syndrome and parental factors (e.g., education). COST-EFFECTIVINESS ANALYSIS/BIA An economic evaluation is performed with the incorporation of medical costs and costs due to loss of productivity for the parents. A detailed costs-study is done for medical specialist care, surgical costs, hospitalization and other costs directly associated with the interventions. Cost prizes of surgery will be determined by the bottom-up micro-costing method. Cost-utility will be measured with QALY (based on EQ-5D utility score) gained, with confidence ellipses and acceptability curves. The impact of conservative policy versus surgery will be investigated on assurance perspective and central level. From the viewpoint of the (health care) government, a societal perspective and perspective of the "budgettair kader zorg" will be highlighted. We will provide a valid framework with budget consequences by a range of predictions. Sensitivity analysis is done.

TIME SCHEDULE Inclusion between Sept 2022 and Sept 2030. Analysis and reporting for each outcome parameter related to age is distributed from January 2025 to September 2031. New recommendation for treatment of trigonocephaly in guideline ready in 2031.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of trigonocephaly

Exclusion Criteria:

* metopic ridge (physiologic early closure of metopic suture)

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with mild, moderate or severe trigonocephaly, between 0 and 8 years of age, excluding metopic ridge (i.e. physiologic early closure of metopic suture).
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2031-02-28 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Head growth | from 0 to 8 years old
  Annual measurement of head circumference in SD for gender and age. Decline in head growth may indicate raised intracranial pressure

SECONDARY OUTCOMES:
fundoscopy | from 1 to 4 years old
  Annual screening for presence of papilledema as sign of raised intracranial pressure
Cognition and behavior | at 0, 2, 4 and 8 years old
  Validated tests for cognition and behavior of the child
refraction and vision | at 1, 4 and 8 years old
  tests taken by orthoptist
forehead shape | at 0, 2, 4, 6 and 8 years old
  3D photos (objective) and VAS score by parents (subjective) to grade the forehead shape
Quality of life and post-traumatic stress | at 0, 2, 4, 6 and 8 years old
  Validated tests to measure quality of life of the child and parents and presence of PTS in parents
Decisional conflict | at 8 years old
  questionnaire to determine whether or not parents are still content with their decision on type of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Irene MJ Mathijssen, MD, PhD, MBA-H, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, ROTTERDAM, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cornelissen MJ, Loudon SE, van Doorn FEC, Muller RPM, van Veelen MC, Mathijssen IMJ. Very Low Prevalence of Intracranial Hypertension in Trigonocephaly. Plast Reconstr Surg. 2017 Jan;139(1):97e-104e. doi: 10.1097/PRS.0000000000002866. PMID 28027242
- [Background] de Planque CA, Petr J, Gaillard L, Mutsaerts HJMM, van Veelen MC, Versnel SL, Dremmen MHG, Mathijssen IMJ. Cerebral Blood Flow of the Frontal Lobe in Untreated Children with Trigonocephaly versus Healthy Controls: An Arterial Spin Labeling Study. Plast Reconstr Surg. 2022 Apr 1;149(4):931-937. doi: 10.1097/PRS.0000000000008931. PMID 35171857
- [Background] Mathijssen IMJ; Working Group Guideline Craniosynostosis. Updated Guideline on Treatment and Management of Craniosynostosis. J Craniofac Surg. 2021 Jan-Feb 01;32(1):371-450. doi: 10.1097/SCS.0000000000007035. No abstract available. PMID 33156164
- [Background] Abdel-Alim T, Iping R, Wolvius EB, Mathijssen IMJ, Dirven CMF, Niessen WJ, van Veelen MC, Roshchupkin GV. Three-Dimensional Stereophotogrammetry in the Evaluation of Craniosynostosis: Current and Potential Use Cases. J Craniofac Surg. 2021 May 1;32(3):956-963. doi: 10.1097/SCS.0000000000007379. PMID 33405445
- [Derived] Tio P, van Staalduinen M, Okkerse J, Dulfer K, Erler N, Loudon S, Telleman M, Abdel-Alim T, Roshchupkin G, Heemskerk S, Polinder S, van Veelen ML, Bannink N, van Driel A, Faasse M, Ista E, Joosten K, Spoor J, Weissbach E, Kats J, Versnel SL, Pleumeekers M, Mathijssen I. Comparing effectiveness of conservative policy to craniofacial surgery in children with metopic synostosis: protocol for an observational cohort study on clinical outcomes, psychosocial well-being and costs in a Dutch academic hospital. BMJ Open. 2025 May 6;15(5):e094112. doi: 10.1136/bmjopen-2024-094112. PMID 40335143